CLINICAL TRIAL: NCT07073768
Title: Comparison Between Efficacy of Trelagliptin and Sitagliptin in Type II Diabetic Patients
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Khyber Medical College, Peshawar (Other)
Responsible Party: Principal Investigator, Dr Aliena Badshah, Assistant Professor of Medicine, Khyber Medical College, Peshawar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KhyberMC
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus Type 2; Glycemic Control for Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; T2DM; Diabetes; Trelagliptin; SYR-472; Sitagliptin; DPP-4 Inhibitors; Dipeptidyl Peptidase-4 Inhibitors; RCT
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — trelagliptin; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trelagliptin Arm (Experimental): A total of 63 participants will receive Trelagliptin 100 mg taken orally once weekly for 3 months. All participants will continue their background metformin therapy as previously prescribed. The study will assess changes in HbA1c, fasting blood sugar, postprandial blood sugar, treatment adherence, and patient satisfaction compared to Sitagliptin.
  Interventions: Drug: Trelagliptin 100 mg
- Sitagliptin Arm (Active Comparator): A total of 63 participants will receive Sitagliptin 100 mg taken orally once daily for 3 months. All participants will continue their background metformin therapy as previously prescribed. The study will assess changes in HbA1c, fasting blood sugar, postprandial blood sugar, treatment adherence, and patient satisfaction compared to Trelagliptin.
  Interventions: Drug: Sitagliptin 100mg OD

INTERVENTIONS:
Drug: Trelagliptin 100 mg — Trelagliptin will be administered as oral tablets at a dose of 100 mg once weekly for 3 months. Participants will continue background metformin therapy as prescribed. Trelagliptin is a dipeptidyl peptidase-4 (DPP-4) inhibitor indicated for type 2 diabetes mellitus and differs from daily DPP-4 inhibitors due to its longer duration of action, allowing weekly dosing.
  Other Names: SYR-472
  Arms: Trelagliptin Arm
Drug: Sitagliptin 100mg OD — Sitagliptin will be administered as oral tablets at a dose of 100 mg once daily for 3 months. Participants will continue background metformin therapy as prescribed. Sitagliptin is a dipeptidyl peptidase-4 (DPP-4) inhibitor indicated for type 2 diabetes mellitus and requires daily dosing.
  Arms: Sitagliptin Arm

SUMMARY:
The goal of this clinical trial is to find out if a medicine called Trelagliptin works as well as another medicine called Sitagliptin to lower blood sugar levels in people with type 2 diabetes who have not reached their target sugar levels with metformin alone.

The main questions this study aims to answer are:

Does Trelagliptin lower average blood sugar levels (measured by HbA1c) as well as Sitagliptin over 3 months? Does Trelagliptin help reduce swings in blood sugar levels compared to Sitagliptin? Are people more likely to stick to taking Trelagliptin, which is taken once a week, than Sitagliptin, which is taken every day? How satisfied are people with their treatment when using Trelagliptin versus Sitagliptin?

Researchers will compare two groups:

One group will take Trelagliptin once a week for 3 months. The other group will take Sitagliptin once a day for 3 months.

Participants in the study will:

Answer questions about their health and how they feel about their diabetes treatment.

Have blood tests to measure blood sugar levels, including:

HbA1c (an average measure of blood sugar over 2-3 months) Fasting blood sugar levels Blood sugar levels two hours after breakfast Keep records of how often they take their medicine.

People can take part in this study if:

They have type 2 diabetes and are taking metformin but still have higher-than-desired blood sugar levels.

They are between certain blood sugar ranges (HbA1c higher than 6.5% but lower than 10%).

They are willing to give informed consent and follow study instructions.

People cannot take part if:

They have type 1 diabetes. They have certain serious health conditions, such as severe kidney disease, heart problems, cancer, or are pregnant.

They are already taking Trelagliptin or are in another clinical study. The study will take place at Khyber Teaching Hospital in Pakistan and will last about 3 months for each participant.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a chronic metabolic disorder associated with significant microvascular and macrovascular complications. In many patients, blood sugar levels remain above target despite treatment with metformin, which is the usual first-line therapy. Additional treatments are often required to achieve optimal glycemic control.

Dipeptidyl peptidase-4 (DPP-4) inhibitors are oral medications used in managing T2DM. They work by preventing the breakdown of incretin hormones, which help regulate insulin secretion and lower blood glucose levels. Most DPP-4 inhibitors, including sitagliptin, require daily dosing. Trelagliptin is a once-weekly DPP-4 inhibitor that has shown higher potency against the DPP-4 enzyme in preclinical and clinical studies. Trelagliptin is approved for use in Japan but has limited availability and data in other countries, including Pakistan.

This randomized controlled trial aims to compare the efficacy and patient experience of Trelagliptin and Sitagliptin in patients with T2DM who have not achieved glycemic targets with metformin alone. The study seeks to evaluate whether once-weekly Trelagliptin provides similar or superior glycemic control compared to once-daily Sitagliptin and whether it improves treatment adherence and patient satisfaction due to reduced dosing frequency.

Participants will be randomly assigned in a 1:1 ratio to either the Trelagliptin group or the Sitagliptin group. The Trelagliptin group will receive a once-weekly dose of 100 mg oral Trelagliptin for 3 months. The Sitagliptin group will receive 100 mg of oral Sitagliptin once daily for 3 months. Both groups will continue metformin therapy as previously prescribed.

Glycemic control will be assessed through measurements of HbA1c at baseline and after 3 months of treatment. Additional evaluations include fasting blood sugar (FBS) and two-hour post-breakfast random blood sugar (RBS) levels measured monthly. Participants will be asked to maintain a medication diary to record doses taken. Treatment adherence will be assessed through the diary entries and through participant interviews. Treatment satisfaction will be evaluated using the Diabetes Treatment Satisfaction Questionnaire (DTSQ).

The study will be conducted at the Department of Medicine, Khyber Teaching Hospital, Pakistan. Data will be collected and analyzed using standard statistical methods. The primary outcome is the change in HbA1c from baseline to 3 months. Secondary outcomes include changes in FBS and RBS levels, treatment adherence rates, and patient-reported treatment satisfaction.

This study is expected to generate valuable evidence on the efficacy and patient acceptability of Trelagliptin in a Pakistani population and may help inform clinical decision-making regarding once-weekly versus daily DPP-4 inhibitor therapy for T2DM.

ELIGIBILITY:
Inclusion Criteria:

* • Type 2 Diabetic patients visiting Medical OPD

  * Patients already maintaining lifestyle modifications and on metformin monotherapy, but not achieving target HbA1c levels.
  * Patients who require treatment with a DPP-4 inhibitors
  * Patients with baseline HbA1c > 6.5% and < 10%
  * Patients willing to provide written informed consent prior to recruitment

Exclusion Criteria:

* • Type 1 Diabetic Patients

  * Patients already using Trelagliptin for type 2 diabetes
  * Patients with severe renal impairment (eGFR < 30ml/min/1.73m2 or on dialysis)
  * Patients with Serious Heart disease or Cerebrovascular disease
  * Patients with Serious Pancreatic or blood disease
  * Patients with malignancy
  * Patients with history of hypersensitivity to DPP-4 inhibitors
  * Patients with history of gastrointestinal resection
  * Pregnant, Breast feeding or planning to be pregnant patients
  * Patients participating in other clinical studies
  * Patients assessed as ineligible by researchers due to any other reason

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-26 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) | 3 Months
  The mean change in HbA1c levels from baseline to 3 months of treatment, comparing Trelagliptin and Sitagliptin groups. HbA1c is measured as a percentage and reflects average blood glucose over the prior 2-3 months.

SECONDARY OUTCOMES:
Change in Fasting Blood Sugar (FBS) | Baseline, monthly for 3 months
  The mean change in fasting blood glucose levels from baseline to monthly time points during 3 months of treatment, comparing Trelagliptin and Sitagliptin groups.
Change in 2-Hour Post-Breakfast Random Blood Sugar (RBS) | Baseline, monthly for 3 months
  The mean change in blood glucose levels measured 2 hours after breakfast, from baseline to monthly time points during 3 months of treatment, comparing Trelagliptin and Sitagliptin groups.

OTHER OUTCOMES:
Treatment Adherence | Throughout 3 months of treatment
  The proportion of prescribed doses taken over the 3-month treatment period, assessed via patient diaries and direct questioning. Reported as a percentage of prescribed doses taken.
Patient Treatment Satisfaction | At 3 months
  Patient-reported satisfaction with treatment as measured by the Diabetes Treatment Satisfaction Questionnaire (DTSQ). Scores will assess satisfaction, convenience, and perceived effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Aliena Badshah, MBBS, FCPS, MRCP, Principal Investigator — Khyber Teaching Hospital
Locations (1):
- Khyber Teaching Hospital / Khyber Medical College, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding sharing individual participant data (IPD) has not yet been made. Considerations include participant privacy, institutional policies, and regulatory requirements.

REFERENCES:
- [Background] Inagaki N, Sano H, Seki Y, Kuroda S, Kaku K. Efficacy and safety of once-weekly oral trelagliptin switched from once-daily dipeptidyl peptidase-4 inhibitor in patients with type 2 diabetes mellitus: An open-label, phase 3 exploratory study. J Diabetes Investig. 2018 Mar;9(2):354-359. doi: 10.1111/jdi.12730. Epub 2017 Oct 30. PMID 28836351
- [Background] Dutta D, Mohindra R, Surana V, Sharma M. Safety and efficacy of once weekly dipeptidyl-peptidase-4 inhibitor trelagliptin in type-2 diabetes: A meta-analysis. Diabetes Metab Syndr. 2022 Apr;16(4):102469. doi: 10.1016/j.dsx.2022.102469. Epub 2022 Mar 21. PMID 35344848
- [Background] Diachenko SS. [Development of medical microbiology in the Ukraine]. Vrach Delo. 1988 May;(5):116-20. No abstract available. Russian. PMID 3047982
- [Background] Deacon CF, Lebovitz HE. Comparative review of dipeptidyl peptidase-4 inhibitors and sulphonylureas. Diabetes Obes Metab. 2016 Apr;18(4):333-47. doi: 10.1111/dom.12610. Epub 2016 Jan 8. PMID 26597596
- [Background] Kim HJ, Kim YS, Lee CB, Choi MG, Chang HJ, Kim SK, Yu JM, Kim TH, Lee JH, Ahn KJ, Min KW, Kyung EJ, Kim YK, Lee KW. Efficacy and Safety of Switching to Teneligliptin in Patients with Type 2 Diabetes Inadequately Controlled with Dipeptidyl Peptidase-4 Inhibitors: 52-Week Results from a Prospective Observational Study. Diabetes Ther. 2021 Nov;12(11):2907-2920. doi: 10.1007/s13300-021-01148-1. Epub 2021 Sep 18. PMID 34536208
- [Background] Stratton IM, Adler AI, Neil HA, Matthews DR, Manley SE, Cull CA, Hadden D, Turner RC, Holman RR. Association of glycaemia with macrovascular and microvascular complications of type 2 diabetes (UKPDS 35): prospective observational study. BMJ. 2000 Aug 12;321(7258):405-12. doi: 10.1136/bmj.321.7258.405. PMID 10938048
- [Background] Grimshaw CE, Jennings A, Kamran R, Ueno H, Nishigaki N, Kosaka T, Tani A, Sano H, Kinugawa Y, Koumura E, Shi L, Takeuchi K. Trelagliptin (SYR-472, Zafatek), Novel Once-Weekly Treatment for Type 2 Diabetes, Inhibits Dipeptidyl Peptidase-4 (DPP-4) via a Non-Covalent Mechanism. PLoS One. 2016 Jun 21;11(6):e0157509. doi: 10.1371/journal.pone.0157509. eCollection 2016. PMID 27328054
- [Background] Glenn JK, Hofmeister RW, Neikirk H, Wright H. Continuity of care in the referral process: an analysis of family physicians' expectations of consultants. J Fam Pract. 1983 Feb;16(2):329-34. PMID 6822803
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC6822803/